CLINICAL TRIAL: NCT01462084
Title: Effectiveness of Adaptive Servoventilation (ASV) in Patients With Central Sleep Apnea Due to Chronic Opioid Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MA-01-10
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea; Central Sleep Apnea (Diagnosis); Chronic Opioid Use
Keywords: sleeping; opioid medications; positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Adaptive Servo-Ventilation (ASV) then BiLevel PAP (Experimental): Adaptive servo-ventilation (ASV) is a form of positive airway pressure (PAP) that is delivered based on the needs of the individual. ASV adjusts to the breathing events the individual is experiencing and provides enough PAP to resolve the breathing event. This is a crossover study, so all patients enter both treatment groups.
  Interventions: Device: Adaptive servo-ventilation (ASV); Device: Bi-Level PAP
- Bi-Level PAP then Adaptive Servo-Ventilation (ASV) (Experimental): Bi-level pressure delivers two pressures, IPAP and EPAP. Both pressures are fixed and do not adjust based on the individuals breathing events. This is a crossover study, so all patients enter both treatment groups.
  Interventions: Device: Adaptive servo-ventilation (ASV); Device: Bi-Level PAP

INTERVENTIONS:
Device: Adaptive servo-ventilation (ASV) — Adaptive servo-ventilation (ASV) is a form of positive airway pressure (PAP) that is delivered based on the needs of the individual.
Device: Bi-Level PAP — Bi-Level PAP delivers therapy at 2 pressures IPAP and EPAP that are fixed.

SUMMARY:
Prospective, randomized, blinded, cross-over study assessing the effectiveness of adaptive servo-ventilation (ASV) in treating patients who have obstructive sleep apnea (OSA) complicated by central sleep apnea (CSA) due to the chronic use of opioid medications

DETAILED DESCRIPTION:
The trial seeks to determine the efficacy and patient comfort of ASV and bi-level positive airway pressure (PAP) modes for the treatment of obstructive sleep apnea (OSA), complicated by CSA secondary to opioid use. Subjects will be randomized to one of two groups, utilizing a cross-over design to evaluate the two modes with the subject as their own control.

Subjects will be asked to undergo two PSG studies; one with ASV titration and one with bi-level treatment, using the current pressure prescription. The study comprises two visits. Subjects will be asked to complete patient satisfaction questionnaires following their PSG studies. It is anticipated that total subject participation will be no longer than one month.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Taking opioid medications for at least 6 months. Opioid medications include but are not limited to: oxycodone, fentanyl, methadone, levorphanol, hydromorphone, and morphine
* Using bi-level PAP for at least 30 days

Exclusion Criteria:

* Primary heart or lung disease, for example: chronic obstructive pulmonary disease, pulmonary fibrosis, severe heart failure, uncorrected congenital heart disease, pulmonary hypertension
* Primary neurologic disease, for example: neuromuscular disease, previous stroke or cognitive impairment
* Narcolepsy
* Acute upper respiratory tract infection
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cao, DO, Principal Investigator — Stanford Center for Human Sleep Research
Locations (1):
- Stanford Center for Human Sleep Research, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from a single sleep center in the United States.
Groups:
- Adaptive Servo-ventilation (ASV): Adaptive servo-ventilation (ASV) is a form of positive airway pressure (PAP) that is delivered based on the needs of the individual. ASV adjusts to the breathing events the individual is experiencing and provides enough PAP to resolve the breathing event. This is a crossover study, so patients in this arm used ASV therapy the first night and then crossed over and used BiLevel PAP the second night.
- Bi-Level PAP: Bi-level PAP delivers two pressures, IPAP and EPAP. Both pressures are fixed and do not adjust based on the individuals breathing events. This is a crossover study, so patients in this arm used Bi-Level PAP therapy the first night and then crossed over and used ASV the second night.
Period: Overall Study
Arm/Group | Adaptive Servo-ventilation (ASV) | Bi-Level PAP
Started | 11 | 10
Included for Analysis | 9 | 9
Completed | 9 | 9
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: A total of 60 patients were screened, 21 met the inclusion criteria, 1 dropped out, 2 patients were not titrated according to protocol and were excluded, leaving data from 18 patients available for inclusion in the analysis.
Groups:
- Overall Study Population: All study patients included in final analysis.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 52.9 [24 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: Subjects completed 2 overnight sleep studies (polysomnography (PSG)). The Apnea Hypopnea Index (AHI) metric is collected from the PSG study. Patients were equally distributed according to the therapy used first (ASV then Bi-Level or Bi-Level then ASV).
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- Adaptive Servo-Ventilation (ASV): All patients received 1 night of therapy using Adaptive servo-ventilation (ASV) and 1 night of therapy using Bi-level PAP. Adaptive servo-ventilation (ASV) is a form of positive airway pressure (PAP) that is delivered based on the needs of the individual. ASV adjusts to the breathing events the individual is experiencing and provides enough PAP to resolve the breathing event. This is a crossover study, so all patients enter both treatment groups.
- Bi-Level PAP: Bi-level pressure delivers two pressures, IPAP and EPAP. Both pressures are fixed and do not adjust based on the individuals breathing events. This is a crossover study, so all patients enter both treatment groups.
Arm/Group | Adaptive Servo-Ventilation (ASV) | Bi-Level PAP
Number analyzed (Participants) | 18 | 18
events/hour | 2.5 (3.5) | 16.3 (20.9)

2. Secondary Outcome: Patient Comfort
Description: Subjects completed patient-satisfaction questionnaires after each polysomnography (PSG) study. Satisfaction with PAP: 0=Very Dissatisfied, 100=Very Satisfied
Time Frame: Up to 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adaptive Servo-ventilation (ASV): Adaptive servo-ventilation (ASV) is a form of positive airway pressure (PAP) that is delivered based on the needs of the individual. ASV adjusts to the breathing events the individual is experiencing and provides enough PAP to resolve the breathing event. Both pressures are fixed and do not adjust based on the individuals breathing events.
Arm/Group | Adaptive Servo-ventilation (ASV) | Bi-Level PAP
Number analyzed (Participants) | 18 | 18
units on a scale | 76.0 (27.2) | 67.8 (28.0)

ADVERSE EVENTS:
Time Frame: Full study duration.
Groups:
- Adaptive Servo-Ventilation (ASV): Adaptive servo-ventilation (ASV) is a form of positive airway pressure (PAP) that is delivered based on the needs of the individual. ASV adjusts to the breathing events the individual is experiencing and provides enough PAP to resolve the breathing event. This is a crossover study, so all patients enter both treatment groups.
Arm/Group | Adaptive Servo-Ventilation (ASV) | Bi-Level PAP
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days